CLINICAL TRIAL: NCT07222540
Title: Expanded Access Program Evaluating SkinTE in the Treatment of Wagner 1 Diabetic Foot Ulcers
Status: Temporarily not available | Type: Expanded Access
Sponsor: PolarityTE (Industry)
Responsible Party: Sponsor
Other Study IDs: PolarityBio EAP - DFU 01
Record Dates: First submitted 2025-10-27; First posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: DFU; Neuropathic Diabetic Ulcer - Foot; Diabetic Foot Disease
Keywords: DFU; PolarityBio; SkinTE

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Biological: SkinTE — SkinTE is an Autologous Heterogeneous Skin Construct (AHSC), which is manufactured from a small piece of healthy full-thickness skin harvested from the patient at the time of randomization to the SkinTE arm. SkinTE is manufactured aseptically by PolarityBio following current Good Manufacturing Practice (cGMP). SkinTE is not cultured ex vivo; rather, it is returned to the provider expeditiously to maintain cellular viability. SkinTE contains multicellular aggregates that contain different types of skin cells, such as keratinocytes, dermal fibroblasts, dermal endothelial cells, and follicular cells, as well as extracellular matrix. The multicellular aggregates have a surface area-to-volume ratio for improved sustenance by imbibition prior to engraftment.
  Other Names: Autologous Heterogeneous Skin Construct

SUMMARY:
The purpose of this EAP is to provide access to SkinTE® for patients with Wagner I Diabetic Foot Ulcers (DFUs). SkinTE® is an autologous investigational product created from a healthy full-thickness skin harvest. SkinTE is applied directly to the wound with the goal of promoting healing.

In addition to providing treatment, the program will collect safety and efficacy data. This data will help us understand the potential risks and benefits of SkinTE® when used in a real-world setting. PolarityBio® provides research funding to the study site to support data collection.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age
2. Subjects are medically optimized with a documented history of Type I or Type II Diabetes Mellitus requiring insulin and/or oral therapy.
3. Presence of a DFU Wagner 1 grade wound on any aspect of the foot, provided that if the malleolus is involved, not more than 50% of the wound is above the mid-point of the medial malleolus. Note: Index Ulcer must maintain Wagner grade 1 from screening to harvest procedure.
4. Index ulcer (i.e., current episode of ulceration) has been present for ≥ four weeks (≥ 28 days) prior to the initial screening visit.
5. If other wound(s) are present on the same foot, they must be more than 2 cm distant from the index ulcer.
6. Ulcer size between 1.0 cm² and 25 cm² post-debridement at screening and day of Harvest, which may occur 3 to 30 days after screening.
7. Adequate circulation to the affected foot documented by a dorsal transcutaneous oxygen measurement (TCOM) or skin perfusion pressure (SPP) measurement of ≥ 30 mmHg, or an Ankle Branchial Index (ABI) of ≥ 0.7 and ≤ 1.2 or Arterial Doppler with a minimum of biphasic flow or Toe Brachial Index (TBI) ≥ 0.75 using the affected study extremity within 30 days of the screening visit.
8. Index ulcer and/or index ulcer limb may have had prior infection(s), but infection(s) must be adequately treated and controlled as defined by IDSA Guidelines PEDIS Grade level 1.
9. The subject can comply with study visits, wound management, and follow-up regimen.
10. The treating investigator has determined that no suitable alternative therapy is available to adequately address the patient's medical needs.
11. Based on the treating investigator's clinical judgment and the severity of the patient's condition, the patient has the potential to derive meaningful benefits from the use of SkinTE.
12. Females of childbearing potential must agree to use effective methods of contraception (birth control pills, barriers, or abstinence) (Screening through End of Study (EOS) and undergo pregnancy tests.
13. Negative pregnancy test for females of childbearing potential (e.g., not post- menopausal for at least one year or surgically sterile).
14. Properly obtained written informed consent.
15. Subjects who previously received SkinTE as part of a prior SkinTE-related trial may be considered for participation, provided a new index ulcer is selected for treatment on the contralateral limb and sponsor approval is granted.

Exclusion Criteria:

1. Participation in another investigational drug or therapeutic device trial within 30 days prior to screening.
2. Use of prohibited medication(s) as defined in this protocol.
3. Presence of diabetes with poor metabolic control, defined as a documented historical HbA1c ≥12.0% within 90 days prior to screening.
4. Subjects with a history of more than two weeks of treatment with immunosuppressants (including systemic corticosteroids > 10mg prednisone (or equivalent) daily dose), or cytotoxic chemotherapy prior to screening.
5. Index ulcer treated within 30 days of screening with prohibited treatment as defined in this protocol.
6. Subjects with presence of gangrene, unstable ischemia, or active Charcot's foot.
7. Subjects with recent lower extremity revascularization within ≤30 days of screening.
8. Based on the treating investigators clinical judgement there is no suspicion of malignancy in the index ulcer.
9. History of osteomyelitis, cellulitis, or other soft tissue infections involving the index ulcer within 30 days of screening.
10. Subjects with exposed internal fixation on the same limb as the index ulcer. [Note: External fixation is allowed if deemed stable by principal investigator.]
11. Active infection of the index ulcer (as defined by IDSA PEDIS Grade 1 guidelines) of the affected limb.
12. History of radiation therapy on the affected limb.
13. Subject is pregnant or breastfeeding.

Sex: All
Age Groups: Child, Adult, Older Adult

REFERENCES:
- [Result] Armstrong DG, Orgill DP, Galiano R, Glat PM, Didomenico L, Sopko NA, Swanson EW, Sigal F, Snyder R, Li WW, Carter M, Zelen CM. A multicenter, randomized controlled clinical trial evaluating the effects of a novel autologous heterogeneous skin construct in the treatment of Wagner one diabetic foot ulcers: Final analysis. Int Wound J. 2023 Dec;20(10):4083-4096. doi: 10.1111/iwj.14301. Epub 2023 Jul 4. PMID 37402533
- [Result] Armstrong DG, Orgill DP, Galiano R, Glat PM, Carter M, Zelen CM, Li WW. Complete wound closure following a single topical application of a novel autologous homologous skin construct: first evaluation in an open-label, single-arm feasibility study in diabetic foot ulcers. Int Wound J. 2020 Oct;17(5):1366-1375. doi: 10.1111/iwj.13404. Epub 2020 May 26. PMID 32453512